CLINICAL TRIAL: NCT02548247
Title: Effect of Consumption of Inulin on Bowel Motor Function in Subjects With Constipation
Brief Title: Effect of Consumption of Orafti® Inulin on Bowel Motor Function in Subjects With Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beneo GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTS528_10
Record Dates: First submitted 2015-09-04; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Healthy; Constipation
Keywords: Stool frequency; Bowel motor function; Orafti® Inulin; Dietary Fiber
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orafti® Inulin (Experimental): Daily consumption of 12g Orafti® Inulin (3x 4g/d) over a period of 4 weeks
  Interventions: Dietary Supplement: Orafti® Inulin
- Placebo (Placebo Comparator): Daily consumption of 12g/ Maltodextrin (3x 4g/d) over a period of 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Orafti® Inulin — Dietary fiber
  Arms: Orafti® Inulin
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
Investigation of the effects of a four week daily consumption of Orafti® Inulin on bowel motor function in subjects with constipation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers without clinical diagnosed diseases with relevant effect on the gastrointestinal system or on visceral motility.
* Constipation defined as an average of 2-3 stools per week. Volunteers should have had constipation for at least the previous 6 months.
* Age ≥ 20 and ≤ 75

Exclusion Criteria:

* Subject under prescription for medication for digestive symptoms such as antispasmodic, laxatives, anti-diarrheic drugs or other digestive auxiliaries.
* Relevant history, presence of any medical disorder or chronic intake of medication/dietary supplements potentially interfering with this trial.
* Subjects with stool frequency of <1 stool every 7 days or more than 3 stools per week.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Stool frequency determined by daily questionnaire | 4 weeks
  Stool frequency determined by daily questionnaire.

SECONDARY OUTCOMES:
Stool consistency rated according to the Bristol Stool Form Scale | 4 weeks
  Stool consistency rated according to the Bristol Stool Form Scale from Type 1 to Type 7.
Questionnaire on Gastrointestinal characteristics | 4 weeks
  Sensation of straining, abdominal discomfort, bloating/distension, passage of gas and feeling of incomplete emptying rated on a 5-point scale (0 = not at all, 1 = very slightly, 2 = slightly, 3 = moderately, 4 = extremely).
Questionnaire on Participant Assessment of Constipation Quality of Life (PAC-QoL) | 4 weeks
  Severity of each symptom rated on a five-point scale from 0 (not at all / none of the time) to 4 (extremely / all of the time).
Faecal microbiota composition determined by illumina sequencing | 4 weeks
  Determined by illumina sequencing.
Stool metabolite profiling determined by GC/LC-MS | 4 weeks
  Determined by GC/LC-MS.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Menzel, MD, Principal Investigator — BioTeSys GmbH
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany

REFERENCES:
- [Derived] Vandeputte D, Falony G, Vieira-Silva S, Wang J, Sailer M, Theis S, Verbeke K, Raes J. Prebiotic inulin-type fructans induce specific changes in the human gut microbiota. Gut. 2017 Nov;66(11):1968-1974. doi: 10.1136/gutjnl-2016-313271. Epub 2017 Feb 17. PMID 28213610
- [Derived] Micka A, Siepelmeyer A, Holz A, Theis S, Schon C. Effect of consumption of chicory inulin on bowel function in healthy subjects with constipation: a randomized, double-blind, placebo-controlled trial. Int J Food Sci Nutr. 2017 Feb;68(1):82-89. doi: 10.1080/09637486.2016.1212819. Epub 2016 Aug 5. PMID 27492975